CLINICAL TRIAL: NCT04858750
Title: Comparison and Evaluation of USSQ (Ureteral Stent Symptom Questionnaire）, OABSS (Overactive Bladder Symptom Score), and the Drainage/Anti-reflux Effect Between Three Kinds of Ureteral D-J（Double-J) Stents in Patients Who Underwent URL (Ureteroscopic Holmium Laser Lithotripsy）
Brief Title: Comparison and Evaluation of USSQ, OABSS, and the Drainage/Anti-reflux Effect Between Three Kinds of Ureteral D-J Stents in Patients Who Underwent URL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XHEC-C-2021-106-1
Record Dates: First submitted 2021-04-14; First posted 2021-04-26 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Urolithiasis; Overactive Bladder Syndrome
Keywords: USSQ; OABSS; double-J stent; ureteroscopic holmium laser lithotripsy
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cook D-J stent group (Other): Patients randomized to this group received Cook (Limerick, Ireland, USI-626-R) D-J stent.
  Note: USI is an unexpandable acronym.
  Interventions: Device: Placement of ureteral D-J stent after ureteroscopic holmium laser lithotripsy
- KYB anti-reflux D-J stent group (Other): Patients randomized to this group received KYB (Shenzhen, China, 3201162) anti-reflux D-J stent.
  Interventions: Device: Placement of ureteral D-J stent after ureteroscopic holmium laser lithotripsy
- Urovision trigonal D-J stent group (Other): Patients randomized to this group received Urovision (Bad Aibling, Germany, ST-230726) trigonal D-J stent.
  Note: ST is an unexpandable acronym. Aibling is a German region name.
  Interventions: Device: Placement of ureteral D-J stent after ureteroscopic holmium laser lithotripsy

INTERVENTIONS:
Device: Placement of ureteral D-J stent after ureteroscopic holmium laser lithotripsy — During ureteral holmium laser lithotripsy operation, after the stones were fragmented, the D-J stents of three different types were placed, the insertion process are exactly the same.

SUMMARY:
Indwelling double-J ureteral stent (D-J stent) are routinely placed in patients who received ureteroscopic lithotripsy (URL) in Xinhua Hospital Urology Department. At present, three types of D-J stents, namely Cook/Kang Yi Bo(KYB)/Urovisionare are used, and usually removed in the day ward four weeks after surgery. This study intends to randomly divide patients with urolithiasis based on the preoperative OABSS (overactive bladder symptom score) questionnaire into three groups, namely Cook D-J stent group, KYB anti-reflux D-J stent group, Urovision trigonal D-J stent group, with corresponding D-J stent indwelled for 4 weeks respectively. The patient's USSQ ureteral stent symptom questionnaire）scale and OABSS scale were collected at 1 week, 4 weeks (before the removal of D-J stents), and 5 weeks (1 week after removal of D-J stents) after URL operation, and the D-J stents removed from the patients were collected, and their drainage and anti-reflux effects were measured in vitro.

ELIGIBILITY:
Inclusion Criteria:

1. Abdominal CT scanning indicating ureteral stones or kidney stones that are less than 2 cm in diameter, and patients who are planning to undergo URL surgery.
2. Age between 18 and 80 years old and capable of providing written informed consent;
3. In general, the heart, lung, liver and kidney function are in well condition, able to tolerate surgical treatment, and comply with research requirements.

Exclusion Criteria:

1. Before the onset of urolithiasis, the patient has suffered from obvious overactive bladder syndrome, or chronic lower urinary tract infection, or urinary anatomic deformities, or had previously undergone urinary tract plastic surgery.
2. Other severe complications, infections, etc. that the researchers believe may make the subject unsuitable for this study.
3. The patient is not a local resident and insists on returning to his howetown for D-J stent removal after the URL operation（so that we are unable to retrieve the D-J stent and conduct the in vitro experiment）.
4. The patient refuses to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Hematuria, lower urinary tract symptoms and other aspects after placement of D-J stent | 1 week (after URL)
  The patients' symptoms are evaluated by complete USSQ (Ureteral Stent Symptom Questionnaire)
Hematuria, lower urinary tract symptoms and other aspects after placement of D-J stent | 1 week (after URL)
  The patients' symptoms are evaluated by OABSS ( Overactive Bladder Symptom Score) scale.
Hematuria, lower urinary tract symptoms and other aspects after placement of D-J stent | 4 weeks (before removal of D-J stent)
  The patients' symptoms are evaluated by complete USSQ (Ureteral Stent Symptom Questionnaire)
Hematuria, lower urinary tract symptoms and other aspects after placement of D-J stent | 4 weeks (before removal of D-J stent)
  The patients' symptoms are evaluated by OABSS ( Overactive Bladder Symptom Score) scale.
Hematuria, lower urinary tract symptoms and other aspects after placement of D-J stent | 5 weeks (1 week after removal of D-J stent)
  The patients' symptoms are evaluated by complete USSQ (Ureteral Stent Symptom Questionnaire)
Hematuria, lower urinary tract symptoms and other aspects after placement of D-J stent | 5 weeks (1 week after removal of D-J stent)
  The patients' symptoms are evaluated by OABSS ( Overactive Bladder Symptom Score) scale.

SECONDARY OUTCOMES:
Drainage effect of D-J stents after being removed | 4 weeks
  The drainage effect of D-J stents removed from the ureters of patients are measured in vitro under liquid manometer
Anti-reflux effect of D-J stents after being removed | 4 weeks
  The anti-reflux effect of D-J stents removed from the ureters of patients are measured in vitro under liquid manometer

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
There might be other serial studies after this study, so we haven't decided yet.